CLINICAL TRIAL: NCT02318979
Title: What is the Optimal Stiffness and Height of a Running-specific Prosthesis?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: W81XWH-11-2-0222
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-05

CONDITIONS: Amputation, Traumatic; Traumatic Amputation of Lower Extremity; Wounds and Injuries
MeSH Terms: conditions — Amputation, Traumatic; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: 10 athletes with a unilateral and 5 athletes with bilateral transtibial amputations used 15 different running-specific prosthetic configurations while they ran at one speed and we measured metabolic rates and biomechanics. 10 athletes with a unilateral and 5 athletes with bilateral transtibial amputations used 15 different running-specific prosthetic configurations while they ran at multiple speeds and we measured top speeds and biomechanics.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Running (Experimental): Participants will run on an instrumented treadmill at one speed using three different prostheses.
  Interventions: Device: Otto Bock prosthesis; Device: Ossur prosthesis; Device: Freedom Innovations prosthesis
- Sprinting (Experimental): Participants will run on an instrumented treadmill at a range of speeds from a jogging speed up to top speed.
  Interventions: Device: Otto Bock prosthesis; Device: Ossur prosthesis; Device: Freedom Innovations prosthesis

INTERVENTIONS:
Device: Otto Bock prosthesis — Participants will run using the Otto Bock prosthesis at a recommended stiffness and height, one category stiffer than recommended at the recommended height, one category softter than recommended at the recommended height, at the optimal stiffness and 2 cm taller, and at the optimal stiffness and 2 cm shorter.
Device: Ossur prosthesis — Participants will run using the Ossur prosthesis at a recommended stiffness and height, one category stiffer than recommended at the recommended height, one category softter than recommended at the recommended height, at the optimal stiffness and 2 cm taller, and at the optimal stiffness and 2 cm shorter.
Device: Freedom Innovations prosthesis — Participants will run using the Freedom Innovations prosthesis at a recommended stiffness and height, one category stiffer than recommended at the recommended height, one category softter than recommended at the recommended height, at the optimal stiffness and 2 cm taller, and at the optimal stiffness and 2 cm shorter.

SUMMARY:
The proposed study aims to characterize the effects of running-specific leg prosthetic stiffness and height during on performance during running and sprinting to optimize running-specific prosthesis prescription. The investigators will collect biomechanical and metabolic data from participants with unilateral and bilateral below the knee amputations while they run at different speeds on a treadmill. This data will be used to understand the effects of running prostheses. Then, these parameters will be used to develop prosthetic prescription techniques for people with below the knee amputations.

ELIGIBILITY:
Inclusion Criteria:

* bilateral or unilateral transtibial amputation
* at least one year of running experience using running-specific prostheses
* 18-55 years old
* no current problems with their prosthesis or residual limb
* at a K4 Medicare Functional Classification Level

Exclusion Criteria:

* Cardiovascular, pulmonary, or neurological disease or disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alena M Grabowski, PhD, Principal Investigator — VA Eastern Colorado Health Care System
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Running: Participants will run on an instrumented treadmill at one speed using different prostheses.
  Participants will run using the Otto Bock, Ossur and Freedom Innovations prostheses at a recommended stiffness and height, one category stiffer than recommended at the recommended height, one category softter than recommended at the recommended height, at the optimal stiffness and 2 cm taller, and at the optimal stiffness and 2 cm shorter.
- Sprinting: Participants will run on an instrumented treadmill at a range of speeds from a jogging speed up to top speed using different prostheses.
  Participants will run using the Otto Bock, Ossur and Freedom Innovations prostheses at a recommended stiffness and height, one category stiffer than recommended at the recommended height, one category softter than recommended at the recommended height, at the optimal stiffness and 2 cm taller, and at the optimal stiffness and 2 cm shorter.
Period: Overall Study
Arm/Group | Running | Sprinting
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Running | Sprinting | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (6.1) | 28 (5) | 30 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 14 | 15 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30
Height [Mean (Standard Deviation); unit: m] | 1.77 (0.08) | 1.77 (0.12) | 1.77 (0.12)
Weight [Mean (Standard Deviation); unit: kg] | 76.1 (14.1) | 76 (12.4) | 76.1 (14.1)

OUTCOME MEASURES:

1. Primary Outcome: Biomechanics
Description: The investigators will measure stance average vertical ground reaction forces during running and sprinting.
Time Frame: 4-10 days
Population: We hypothesized that prosthetic configurations would affect stance average vertical ground reaction forces.
Measure: Mean (Standard Deviation); unit: N/kg
Arm/Group | Running | Sprinting
Number analyzed (Participants) | 15 | 15
N/kg | 0.1386 (0.0031) | 0.1835 (0.0204)

2. Secondary Outcome: Metabolic Demand
Description: The investigators will measure rates of oxygen consumption and carbon dioxide production during running to determine the optimal prosthesis for each participant.
Time Frame: 4 days
Population: Best metabolic cost for a running-specific prosthetic configuration.
Measure: Mean (Standard Error); unit: Net CoT (J/kg/m)
Groups:
- Running - Unilateral; Running-Bilateral: Participants will run on an instrumented treadmill at one speed using different prostheses.
  Participants will run using the Otto Bock, Ossur and Freedom Innovations prostheses at a recommended stiffness and height, one category stiffer than recommended at the recommended height, one category softter than recommended at the recommended height, at the optimal stiffness and 2 cm taller, and at the optimal stiffness and 2 cm shorter.
Arm/Group | Running - Unilateral | Running-Bilateral
Number analyzed (Participants) | 10 | 5
Net CoT (J/kg/m) | 3.82 (1.5) | 3.38 (1.0)

3. Secondary Outcome: Top Speed
Description: The investigators will measure the top sprinting speed to determine the optimal prosthesis for each participant.
Time Frame: 4-10 days
Population: Fastest top speed for a running-specific prosthetic configuration.
Measure: Mean (Standard Deviation); unit: m/s
Groups:
- Sprinting - Unilateral; Sprinting - Bilateral: Participants will run over a range of speeds up to their top speed on an instrumented treadmill using different prostheses.
  Participants will run using the Otto Bock, Ossur and Freedom Innovations prostheses at a recommended stiffness and height, one category stiffer than recommended at the recommended height, one category softter than recommended at the recommended height, at the optimal stiffness and 2 cm taller, and at the optimal stiffness and 2 cm shorter.
Arm/Group | Sprinting - Unilateral | Sprinting - Bilateral
Number analyzed (Participants) | 10 | 5
m/s | 8.18 (1.00) | 9.42 (0.90)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Running | Sprinting
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-30): https://cdn.clinicaltrials.gov/large-docs/79/NCT02318979/Prot_SAP_000.pdf